CLINICAL TRIAL: NCT03132207
Title: The 4th Month Oral Consultation at Pregnant Women : Investigation Carried in Pregnant Women and Health Care Professionals of Nantes and Brest
Brief Title: The 4th Month Oral Consultation at Pregnant Women
Acronym: C4M
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Université de Nantes (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0138
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Periodontal Diseases; Pregnancy
Keywords: Oral Health; Pregnancy; Prevention; adverse pregnancy outcomes
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women: Pregnant women attending hospital during pregnancy monitoring and / or being hospitalized in one of the maternity wards associated with the project.
  Interventions: Other: Non interventionel study
- Professional: health professionals in charge of the follow-up of these pregnant women and their childbirth.
  Interventions: Other: Non interventionel study

INTERVENTIONS:
Other: Non interventionel study — Only one questionnaire will be done for women and professional

SUMMARY:
Epidemiological studies have suggested that maternal periodontitis affects the fetal-placental unit, with an increased risk of adverse pregnancy outcome. Indeed, it has been suggested that the direct or indirect action of parodontopathogenic bacteria induces an inflammatory cascade that leads to spontaneous premature labor. Also, non-treatment of caries and periodontal disease can lead to acute pain and stress. This may promote self-medication and the inappropriate use of analgesic medications, potentially harmful to the health of the fetus. As part of the prevention of complications of pregnancy associated with oral diseases, the National Agency for Accreditation and Evaluation in Health (ANAES) has set up a system that allows any pregnant woman to consult between the 4th and 7th month of pregnancy, an oral health professional to carry out a complete assessment and free care. This study aims at evaluating this device among pregnant women and healthcare professionals 4 years after its implementation. On the other hand, it will make it possible to look for a possible link between the realization of an oral prenatal follow-up and the outcome of the pregnancy.

DETAILED DESCRIPTION:
This study will concern two populations:

* pregnant women attending hospital during pregnancy monitoring and / or being hospitalized in one of the maternity wards associated with the project,
* health professionals in charge of the follow-up of these pregnant women and their childbirth.

The study will include:

* 500 pregnant women: 300 in Nantes and 200 in Brest
* 150 health professionals.

ELIGIBILITY:
Inclusion Criteria for pregnant women:

Any woman who is consulting or hospitalized in a maternity unit participating in the project is eligible for the following criteria:

* a voluntary adult woman who gave oral consent
* pregnant women (2nd and 3rd trimesters) or postpartum women hospitalized at the maternity ward
* women agreeing to participate in the study

For health professionals:

* midwife, maieutician, gynecologist and obstetrician,
* have graduated from a specialty,
* agreeing to participate in the study

Exclusion Criteria for pregnant women:

* child
* person under curatorship, under guardianship, deprived of liberty,
* refuse to fill in the questionnaire,
* no understanding of oral or written French,

For health professionals:

- Not graduated

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will concern two populations:
  * pregnant women attending hospital during pregnancy monitoring and / or being hospitalized in one of the maternity wards associated with the project,
  * health professionals in charge of the follow-up of these pregnant women and their childbirth.
Sampling Method: Non-Probability Sample
Enrollment: 622 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

PRIMARY OUTCOMES:
Evaluate the participation rate of pregnant women in the 4th month oral consultation in Nantes and Brest. | 4th month of pregnancy
  Participation (yes / no) in the oral consultation of the 4th month. This is the answer to question 10 of the patient questionnaire.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Brest University Hospital, Brest
  - Nantes University Hospital, Nantes

IPD SHARING:
Plan to Share IPD: No